CLINICAL TRIAL: NCT04319653
Title: Development of a Pelvic Cavity Characterization Algorithm Through the Acquisition of MRI Images and Pressure Measurement by an Intravaginal Probe
Acronym: MI-IRM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulty
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018_28; 2019-A00560-57 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Floor Disorders
Keywords: Geometrical reconstruction; Pelvic Floor Disorders; FE models; Pelvic system; MRI
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic pelvic MRI (Experimental)
  Interventions: Device: Dynamic pelvic MRI with intravaginal probe with pressure sensor

INTERVENTIONS:
Device: Dynamic pelvic MRI with intravaginal probe with pressure sensor — Dynamic pelvic MRI with intravaginal probe and intravaginal and intrarectal opacification gel

SUMMARY:
The conditions such as childbirth or endometriosis can lead to a change in the mobility of the pelvic organs (bladder, vagina, rectum and uterus). The purpose of the study is to study in a personalized way each woman the characteristics of the tissues of their pelvis and to be able to personalize the treatments (surgery, injection, rehabilitation, etc.). Women requiring pelvic MRI may participate in the study. The pelvic dynamic MRI will be done with an intravaginal probe which will be inserted by the patient herself as well as gel in the anus and vagina which will allow to obtain the data on the characteristics of the pelvic tissues of each woman with a 3D reconstruction.

ELIGIBILITY:
Inclusion Criteria:

All:

* Understanding of the French language
* Signature of informed consent
* Insured social patient

For pregnant women:

* Primiparous women
* with no severe maternal-fetal pathology
* with no scheduled caesarean section at the time of the MRI

For women with prolapse:

- Requires pelvic MRI

Exclusion Criteria:

* Minor
* Person who does not have social security
* Person with ongoing vaginal infection
* Pregnant woman during the first or third trimester of pregnancy
* Pregnant woman with broken water pocket
* Bi-cicatricial uterus
* IVF
* Person wearing a pace maker or any intra-body metal implant (if "tube" MRI)
* Claustrophobic person (if "tube" MRI)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The recruitment of patients will be done during a consultation within the Obstetric Gynecology Department CHU of Lille to select those requiring a pelvic MRI.
Enrollment: 1 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
3D reconstruction of the pelvic cavity | at 1 month
  Characterization of the pelvic cavity through a double assessment: a pelvic MRI sequence and an intravaginal pressure probe.

CONTACTS AND LOCATIONS:
Overall Officials: Michel COSSON, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHU, Lille, France